CLINICAL TRIAL: NCT01339429
Title: Evaluation of the Performance and Safety of a Simplified Negative Pressure Wound Therapy Device
Brief Title: Simplified Negative Pressure Wound Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Center for Integration of Medicine & Innovative Technology (Other); Fogarty International Clinical Research Scholarship (Unknown)
Responsible Party: Principal Investigator, Robert Riviello, Instructor in Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-002279/1
Record Dates: First submitted 2011-03-28; First posted 2011-04-20 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Wounds
Keywords: wound; negative pressure wound therapy; non-powered negative pressure wound therapy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- simplified Negative Pressure Wound Therapy (Experimental): The simplified Negative Pressure device will be placed on subjects selected from the hospital ward and meeting the eligibility criteria.
  Interventions: Device: simplified negative pressure wound therapy device (Wound Pump device)

INTERVENTIONS:
Device: simplified negative pressure wound therapy device (Wound Pump device) — A non-powered negative pressure device utilizing a bellows attached to a specialized dressing via drainage tube to promote healing of open wounds.
  Other Names: Wound Pump, manufactured by Worldwide Innovative Healthcare, Inc.

SUMMARY:
The objective of this study is to implement a simplified Negative Pressure Wound Therapy (sNPWT) device in a low resource setting. The investigators hypothesize that the sNPWT device is at least equivalent to commercially available NPWT devices. Therefore, the specific aims of this study will be to measure: 1. the mechanical properties of the sNPWT device and 2. the adverse events associated with the sNPWT device.

ELIGIBILITY:
Inclusion Criteria:

* open wound appropriate for NPWT
* wound size greater than 2 cm2 and less than 150 cm2
* adequate adjacent intact skin for application of sNPWT
* adequate contour of wound location for application of sNPWT
* patient is expected to tolerate change of the NPWT dressing with the chosen analgesia and sedation plan by the treating physician
* the patient is expected to remain clinically stable for the duration of the study
* the patient is to remain hospitalized for the duration of the study
* patient or their legal representative is willing and able to sign an IRB-approved informed consent
* patient less than 21 years old is willing to sign an approved assent form if able to sign

Exclusion Criteria:

* exposed blood vessels
* ischemic wound
* wound with necrotic tissue requiring further debridement at the time of enrollment
* infection
* acute osteomyelitis
* malignancy in the wound
* latex or rubber containing product sensitivity

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riviello, M.D., M.P.H., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- Rwanda (2):
  - Rwinkwavu Hospital, Rwinkwavu, Kayonza District
  - Central University Teaching Hospital in Kigali, Kigali, Kigali

REFERENCES:
- [Derived] Mody GN, Zurovcik DR, Joharifard S, Kansayisa G, Uwimana G, Baganizi E, Ntakiyiruta G, Mugenzi D, Riviello R. Biomechanical and safety testing of a simplified negative-pressure wound therapy device. Plast Reconstr Surg. 2015 Apr;135(4):1140-1146. doi: 10.1097/PRS.0000000000001101. PMID 25502858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital wards were surveyed daily over the study period for eligible patients. Photographs of wounds ranging from 2-150 cm2 in size and clinical histories were reviewed for study enrollment eligibility criteria.
Pre-assignment Details: 47 patients consented. 6 did not meet inclusion criteria. 1 voluntarily withdrew. 4 not enrolled due to clinical changes.
Groups:
- Simplified Negative Pressure Wound Therapy: The simplified negative pressure wound therapy device was placed on subjects selected from hospital wards and meeting the eligibility criteria regarding wound size and condition. Inclusion criteria included age 14 years or older, adequate adjacent intact skin and wound location for application of the sNPWT dressing, adequate pain control, and anticipated clinically stability and hospitalization for the duration of the study. Exclusion criteria were exposed blood vessels, evidence of ischemia, necrotic tissue requiring further debridement, infection, osteomyelitis, and malignancy in the wound.
  Simplified negative pressure wound therapy device: A non-powered negative pressure wound therapy device utilizing a bellows connected to a specialized dressing via a drainage tube.
Period: Overall Study
Arm/Group | Simplified Negative Pressure Wound Therapy
Started | 41
Completed | 37
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Simplified Negative Pressure Wound Therapy: The simplified Negative Pressure device will be placed on subjects selected from the hospital wards and meeting the eligibility criteria.
  simplified Negative Pressure device: A non-powered negative pressure device utilizing a bellows which is compressed every eight hours.
Arm/Group | Simplified Negative Pressure Wound Therapy
Number analyzed (Participants) | 41
Age, Customized [Number; unit: participants]
  14 to 90 Years | 41
Sex/Gender, Customized [Number; unit: participants] — Gender was not consistently recorded.
  participants
    Male | 2
    Female | 2
    Unknown | 37
Region of Enrollment [Number; unit: participants]
  Rwanda | 41

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Negative Pressure
Description: The negative pressure being delivered by the device was measured on a daily basis for three days. Maintenance of negative pressure was defined as negative pressure delivery within 75% of the starting negative pressure amount.
Time Frame: 3 days
Population: 85 dressings were applied. 5 applications excluded due to a change in patient condition, unrelated to sNPWT. 9 dressings excluded due to occlusion of the drainage tube. 71 dressings were analyzed in total.
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: dressings
Groups:
- Simplified Negative Pressure Wound Therapy: The simplified negative pressure wound therapy device will be placed on subjects selected from the surgical ward and meeting the eligibility criteria regarding wound size and condition.
  Simplified negative pressure wound therapy device: A non-powered negative pressure wound therapy device utilizing a bellows connected to a specialized dressing.
Arm/Group | Simplified Negative Pressure Wound Therapy
Number analyzed (Participants) | 37
Number analyzed (dressings) | 71
hours | 22.2 (27.0)

2. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Any adverse events, including bleeding, wound complication, or change in patient condition during the trial period will be recorded.
Time Frame: 3 days
Measure: Number; unit: participants
Units Other Than Participants: dressings
Arm/Group | Simplified Negative Pressure Wound Therapy
Number analyzed (Participants) | 37
Number analyzed (dressings) | 71
participants | 0

ADVERSE EVENTS:
Groups:
- Simplified Negative Pressure Wound Therapy: The simplified negative pressure wound therapy device was placed on subjects selected from the hospital wards and meeting the eligibility criteria regarding wound size and condition.
  Simplified negative pressure wound therapy device: A non-powered negative pressure wound therapy device utilizing a bellows connected to a specialized dressing.
Arm/Group | Simplified Negative Pressure Wound Therapy
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplified Negative Pressure Wound Therapy (N=41)
Fever (Immune system disorders) | 1 (1) — Fever in an immunocompromised patient after discontinuation of the sNPWT device. Deemed not to be serious nor unexpected by IRB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No